CLINICAL TRIAL: NCT01665807
Title: A Time-Motion Study to Compare Self-vaccination With Intanza® Intradermal Influenza Vaccine to Nurse-administered Vaxigrip® Intramuscular Influenza Vaccine in Small Group Settings of Health Care Workers
Brief Title: A Time-motion Study Comparing Self- to Nurse-vaccination With Influenza Vaccine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Brenda Coleman (Other)
Collaborators: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor-Investigator, Brenda Coleman, Clinical Scientist, Mount Sinai Hospital, Canada
Organization: Mount Sinai Hospital, Canada (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: SP1203
Record Dates: First submitted 2012-08-13; First posted 2012-08-15 (Estimated); Results first posted 2013-10-01 (Estimated); Last update posted 2017-04-19 (Actual); Status verified 2017-03

CONDITIONS: Influenza; Vaccination Site Reactions (HT)
Keywords: influenza; vaccine; administration
MeSH Terms: conditions — Influenza, Human | interventions — vaxigrip

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Nurse-administered IM (Experimental): Nurse-administered intramuscular influenza vaccine (Vaxigrip, 0.5 mL)
  Interventions: Biological: Vaxigrip
- Self-administered intradermal (Experimental): Self-administered intradermal influenza vaccine (Intanza 0.1 mL)
  Interventions: Biological: Intanza
- Repeat self-administration intradermal (Active Comparator): Self-administration of intradermal influenza vaccine (Intanza 0.1 mL) by participants who self-administered an intradermal vaccine in our 2010 study
  Interventions: Biological: Intanza

INTERVENTIONS:
Biological: Intanza — Intanza influenza vaccine, trivalent split-virion, inactivated, approved for the 2012-2013 influenza season in northern hemisphere
  Arms: Repeat self-administration intradermal; Self-administered intradermal
Biological: Vaxigrip — Influenza vaccine, trivalent, split-virion, inactivated, approved for the 2012-2013 influenza season in the northern hemisphere
  Arms: Nurse-administered IM

SUMMARY:
The investigators hypothesize that people working in an acute care hospital setting will be able to successfully self-administer the intradermal vaccine (Intanza) in less time than nurse-administration of the regular intramuscular influenza vaccine (Vaxigrip). The investigators also hypothesize that people administering the intradermal vaccine for the second time will take less time to successfully administer than people administering it for the first time.

DETAILED DESCRIPTION:
Vaccination of healthcare workers has been shown to reduce mortality and morbidity in the patients they care for, as well as reducing illness and absenteeism in the healthcare workers themselves, and healthcare worker vaccination programs have been shown to be cost-effective for hospitals because of the reduced absenteeism. Although influenza vaccination programs based on nurse-administered intramuscular vaccination are effective, easy access to vaccination for hospital staff remains a challenge, in part because of large numbers of staff working evening, night and weekend shifts. In addition, in the Canadian setting, increasing the efficiency of all hospital programs is a priority. If regular recipients of seasonal vaccine became accustomed to the practice, self-administration may significantly improve the efficiency of pandemic mass vaccination campaigns.

ELIGIBILITY:
Inclusion Criteria:

* Medically stable men or women 18 to 69 years of age (inclusive)
* Work in any capacity (including physicians and midwives with admitting privileges), volunteer, or student at participating hospital
* Able to read, understand, and respond to questionnaires
* Able to read, understand, and sign an informed consent form
* Available for follow-up for 8 days post-vaccination
* Participants in Part B (repeat administration) of the study must also have participated in the previous randomized control trial of self- versus nurse-administered intradermal influenza vaccine and must have attempted to self-administer the vaccine

Exclusion Criteria:

* Already received 2012-13 influenza vaccine
* History of a severe reaction following influenza vaccination
* Known allergy to components of study vaccines (Intanza® or Vaxigrip®)
* History of Guillain-Barré Syndrome (GBS) within 8 weeks following influenza vaccination
* Acute febrile illness (>37.9ºC orally) within the past 48 hours (participation may be deferred until recovery for these subjects)

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 868 (Actual)
Dates: Start 2012-09; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brenda L Coleman, PhD, Principal Investigator — MOUNT SINAI HOSPITAL; Melissa Barton, Study Director — MOUNT SINAI HOSPITAL; Christine Moore, Study Director — MOUNT SINAI HOSPITAL; Shelly A McNeil, MD, Principal Investigator — Canadian Centre for Vaccinology; Joanne M Langley, MD, Study Director — Canadian Centre for Vaccinology; Scott A Halperin, MD, Study Director — Canadian Centre for Vaccinology; Allison J McGeer, MD, FRCPC, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (2):
- Canada (2):
  - Center for Vaccinology, Halifax, Nova Scotia
  - Mount Sinai Hospital, Toronto, Ontario

REFERENCES:
- [Derived] Coleman BL, McNeil SA, Langley JM, Halperin SA, McGeer AJ. Differences in efficiency, satisfaction and adverse events between self-administered intradermal and nurse-administered intramuscular influenza vaccines in hospital workers. Vaccine. 2015 Nov 27;33(48):6635-40. doi: 10.1016/j.vaccine.2015.10.095. Epub 2015 Oct 31. PMID 26529074

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Sites: 2 acute care hospitals in Canada Dates: September 25, 2012 to November 20, 2012
Pre-assignment Details: People who had self-administered intradermal influenza vaccine in past were only eligible for the "repeat" self-administration arm.
  No other pre-assignment eligibility criteria.
Groups:
- Nurse-administered IM: Nurse-administered intramuscular influenza vaccine (Vaxigrip, 0.5 mL)
  Vaxigrip : Influenza vaccine, trivalent, split-virion, inactivated, approved for the 2012-2013 influenza season in the northern hemisphere
- Repeat Self-administration Intradermal: Self-administration of intradermal influenza vaccine (Intanza 0.1 mL) by participants who self-administered an intradermal vaccine in our 2010 study
  Intanza : Intanza influenza vaccine, trivalent split-virion, inactivated, approved for the 2012-2013 influenza season in northern hemisphere
- Self-administered Intradermal: Self-administered intradermal influenza vaccine (Intanza 0.1 mL)
  Intanza : Intanza influenza vaccine, trivalent split-virion, inactivated, approved for the 2012-2013 influenza season in northern hemisphere
Period: Overall Study
Arm/Group | Nurse-administered IM | Repeat Self-administration Intradermal | Self-administered Intradermal
Started | 411 | 58 | 402
Completed | 409 | 58 | 401
Not Completed | 2 | 0 | 1
Not completed — Withdrawal by Subject | 2 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Repeat Self-administered Intradermal: Self-administration (2) of intradermal influenza vaccine (Intanza 0.1 mL) by participants who self-administered an intradermal vaccine in our 2010 study
  Intanza : Intanza influenza vaccine, trivalent split-virion, inactivated, approved for the 2012-2013 influenza season in northern hemisphere
- Total: Total of all reporting groups
Arm/Group | Nurse-administered IM | Repeat Self-administered Intradermal | Self-administered Intradermal | Total
Number analyzed (Participants) | 411 | 58 | 402 | 871
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 386 | 58 | 391 | 835
  >=65 years | 25 | 0 | 11 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.0 (13.2) | 40.2 (11.3) | 41.2 (12.6) | 42.5 (12.9)
Sex/Gender, Customized [Number; unit: participants]
  Female | 295 | 39 | 282 | 616
  Male | 113 | 19 | 119 | 251
Region of Enrollment [Number; unit: participants]
  Canada | 411 | 58 | 402 | 871

OUTCOME MEASURES:

1. Primary Outcome: Time to Administer Influenza Vaccine (in Seconds)
Description: Time required to explain vaccination, obtain consent, administer vaccine, and register vaccination
Time Frame: Vaccination (Day 0)
Measure: Median (Full Range); unit: seconds
Arm/Group | Nurse-administered IM | Repeat Self-administration Intradermal | Self-administered Intradermal
Number analyzed (Participants) | 408 | 57 | 395
seconds | 90.0 [18.0 to 235.3] | 182.0 [42.5 to 671.1] | 62.6 [29.8 to 97.7]

2. Secondary Outcome: Acceptability of Vaccine
Description: The post-vaccination (Day 0) and follow-up (Day 8) questionnaires include questions on the participant's preference for intradermal or intramuscular injections and questions about their preference for administration by a healthcare provider or self-vaccination.
Time Frame: Follow up (Day 8)
Reporting Status: Not Posted

3. Secondary Outcome: Success Rate
Description: Successful administration, defined as being able to self-vaccinate (or for RN to provide vaccine) on the first attempt. Will be calculated using the number of participants who are successful divided by the number of participants randomized to group.
Time Frame: Vaccination (Day 0)
Measure: Number; unit: participants
Arm/Group | Nurse-administered IM | Repeat Self-administration Intradermal | Self-administered Intradermal
Number analyzed (Participants) | 409 | 58 | 401
participants | 0 | 58 | 394

4. Secondary Outcome: Local & Systemic Reactogenicity
Description: Maximum self-reported diameter of redness, induration, and swelling, and maximum intensity and duration of itchiness, fever, muscle ache, joint pain, headache, fatigue, feeling unwell, and injection site pain as reported on Day 8 after vaccination
Time Frame: Follow up (Day 8)
Reporting Status: Not Posted

5. Secondary Outcome: Pain at Injection Site
Description: Self-perceived pain of injection will be recorded on an 11-point visual analogue scale immediately following vaccination (Day 0) and at follow-up (Day 8)
Time Frame: Follow up (Day 8
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Nurse-administered IM | Repeat Self-administration Intradermal | Self-administered Intradermal
Serious Adverse Events (participants affected / at risk) | 0/409 | 0/58 | 0/401
Other Adverse Events (participants affected / at risk) | 0/409 | 0/58 | 0/401

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No